CLINICAL TRIAL: NCT05816265
Title: Effects of IV Iron Replacement on Exercise Capacity in Individuals With Heart Failure With Reduced Ejection Fraction and Iron Deficiency
Brief Title: Effects of IV Iron Replacement on Exercise Capacity in Individuals With Heart Failure
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Radha Gopalan (Other)
Collaborators: American Regent, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Radha Gopalan, Clinical Professor of Medicine and Cardiology, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001297
Record Dates: First submitted 2023-03-31; First posted 2023-04-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Iron-deficiency
Keywords: Reduced ejection fraction; Exercise; iron supplementation; Cardiopulmonary exercise; peak oxygen uptake
MeSH Terms: conditions — Heart Failure; Anemia, Iron-Deficiency; Motor Activity | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: Randomization will be 1:1 between control group and iron group. Subjects randomized to the iron group will receive iron infusion 1 week after enrollment. The control group will not receive iron replacement infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Iron Infusion Group (Experimental): Subjects will receive iron infusion 1 week after enrollment. Dosage of iron will be at discretion of physicians
  Interventions: Drug: IV Iron Infusion Group
- Control Group (No Intervention): Subjects will not receive iron replacement infusion.

INTERVENTIONS:
Drug: IV Iron Infusion Group — Subjects will receive IV Iron Infusion. Dosage of iron will be at discretion of physicians
  Other Names: Ferric carboxymaltose injection
  Arms: IV Iron Infusion Group

SUMMARY:
Patients with heart failure with reduced ejection fraction and iron deficiency will be randomized to either receive iron infusion or be in the control group. The study is looking at how iron replacement affects exercise capacity as measured by peak oxygen uptake.

DETAILED DESCRIPTION:
Currently 5.7 million people in the United States (US) have Heart Failure and it is expected that by 2030 more than 8 million people will have this condition, accounting for a 46 % increase in prevalence. Iron deficiency and anemia are both common findings in patients with heart failure and contribute to morbidity and mortality. The average cost of hospital admissions for heart failure are about $17,000-25,000; creating a large burden on health-care resources and iron replacement may serve to reduce readmissions at less than a tenth of the cost.

The working hypothesis to support Iron supplementation is that it improves oxygen carrying capacity, thereby improving exercise tolerance. Exercise tolerance in patients with heart failure is an important prognostic indicator.

Role of iron supplementation has been investigated to improve quality of life and outcomes in patients with heart failure and two large multi-centric trails. FAIR-HF and CONFIRM-HF have both showed significant improvement in symptoms and six-minute walk distances in patients with HFrEF after IV iron supplementation. This was found to be true for both anemic and non-anemic patients. Despite the current data, IV iron supplementation is currently only a class IIb recommendation for HFrEF and routine testing of iron studies, is not a part of practice guidelines for heart failure management.

Part of what makes the existing data less compelling is that exercise tolerance was assessed using a 6-minute walk test and though it correlates with functional capacity, it is a sub-maximal exercise test and cannot assess the peak oxygen uptake. Individuals with heart failure are often unable to attain this peak oxygen uptake. The inability to increase O2 uptake with exercise is what affects exercise capacity.

The study aims to bridge the gap between the response seen after IV iron supplementation and the change in physiology we attribute to it using a formal Cardiopulmonary exercise testing. A peak VO2 provides the most objective assessment of functional capacity in patients with HF. This parameter is a surrogate marker for the maximal cardiac output that an individual can achieve. A modest increase in peak VO2 of 6% at 3 months of exercise training has been associated with a reduction in mortality by 5 %.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years
* New York Heart Association Class II-III heart failure
* Left ventricular dysfunction with left ventricular ejection fraction ≤ 40%
* Ferritin < 100 ng/mL or 100-300 ng/mL with transferrin saturation (TSAT) < 20%
* Patients deemed by an attending physician to require intravenous iron therapy
* The patient is willing and able to comply with the protocol and has provided written informed consent

Exclusion Criteria:

* Iron overload disorders or allergy, concomitant nutritional deficiencies- B12 and folate
* Recent Acute Coronary Syndrome
* Physical barriers to exercise capacity
* Currently presenting in heart failure exacerbation
* Declined participation
* Chronic liver disease
* NYHA class IV
* Active bleeding
* Pregnancy
* Life expectancy ≤ 12 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity | 2 months after IV iron infusion
  Cardiopulmonary exercise testing will be administered to measure Peak V02. During the exercise testing a special mouthpiece that can measure oxygen and carbon dioxide is used to measure peak oxygen uptake.
Patient subjective outcome measures | 2 months after IV iron infusion
  Subjects will complete the Kansas City Cardiomyopathy Questionnaire.The lowest score is 0 and the highest score is 100. The higher the score is, the better the quality of life.

SECONDARY OUTCOMES:
Objective Quality of Life measures | 2 months after IV iron infusion
  A 6-minute walk test will be administered to determine if the NYHA class has improved.

CONTACTS AND LOCATIONS:
Locations (1):
- Banner - University Medical Center, Phoenix campus, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Only coded research data will be shared for data analysis by study team. Only limited data set may be shared with sponsor if requested according to data agreement. Future use data will be de-identified and stored in REDCap and only utilized by the investigator's department researchers. Publications and reports will be de-identified.

REFERENCES:
- [Background] Jankowska EA, Rozentryt P, Witkowska A, Nowak J, Hartmann O, Ponikowska B, Borodulin-Nadzieja L, Banasiak W, Polonski L, Filippatos G, McMurray JJ, Anker SD, Ponikowski P. Iron deficiency: an ominous sign in patients with systolic chronic heart failure. Eur Heart J. 2010 Aug;31(15):1872-80. doi: 10.1093/eurheartj/ehq158. Epub 2010 Jun 21. PMID 20570952
- [Background] von Haehling S, Ebner N, Evertz R, Ponikowski P, Anker SD. Iron Deficiency in Heart Failure: An Overview. JACC Heart Fail. 2019 Jan;7(1):36-46. doi: 10.1016/j.jchf.2018.07.015. Epub 2018 Dec 12. PMID 30553903
- [Background] Ebner N, von Haehling S. Iron deficiency in heart failure: a practical guide. Nutrients. 2013 Sep 23;5(9):3730-9. doi: 10.3390/nu5093730. PMID 24064572
- [Background] Anker SD, Comin Colet J, Filippatos G, Willenheimer R, Dickstein K, Drexler H, Luscher TF, Bart B, Banasiak W, Niegowska J, Kirwan BA, Mori C, von Eisenhart Rothe B, Pocock SJ, Poole-Wilson PA, Ponikowski P; FAIR-HF Trial Investigators. Ferric carboxymaltose in patients with heart failure and iron deficiency. N Engl J Med. 2009 Dec 17;361(25):2436-48. doi: 10.1056/NEJMoa0908355. Epub 2009 Nov 17. PMID 19920054
- [Background] Ezekowitz JA, McAlister FA, Armstrong PW. Anemia is common in heart failure and is associated with poor outcomes: insights from a cohort of 12 065 patients with new-onset heart failure. Circulation. 2003 Jan 21;107(2):223-5. doi: 10.1161/01.cir.0000052622.51963.fc. PMID 12538418
- [Background] Klip IT, Comin-Colet J, Voors AA, Ponikowski P, Enjuanes C, Banasiak W, Lok DJ, Rosentryt P, Torrens A, Polonski L, van Veldhuisen DJ, van der Meer P, Jankowska EA. Iron deficiency in chronic heart failure: an international pooled analysis. Am Heart J. 2013 Apr;165(4):575-582.e3. doi: 10.1016/j.ahj.2013.01.017. Epub 2013 Feb 22. PMID 23537975
- [Background] Okonko DO, Mandal AK, Missouris CG, Poole-Wilson PA. Disordered iron homeostasis in chronic heart failure: prevalence, predictors, and relation to anemia, exercise capacity, and survival. J Am Coll Cardiol. 2011 Sep 13;58(12):1241-51. doi: 10.1016/j.jacc.2011.04.040. PMID 21903058
- [Background] Lim EA, Sohn HS, Lee H, Choi SE. Cost-utility of ferric carboxymaltose (Ferinject(R)) for iron-deficiency anemia patients with chronic heart failure in South Korea. Cost Eff Resour Alloc. 2014 Sep 10;12:19. doi: 10.1186/1478-7547-12-19. eCollection 2014. PMID 25278814
- [Background] Wang G, Zhang Z, Ayala C, Wall HK, Fang J. Costs of heart failure-related hospitalizations in patients aged 18 to 64 years. Am J Manag Care. 2010 Oct;16(10):769-76. PMID 20964473
- [Background] Fang J, Mensah GA, Croft JB, Keenan NL. Heart failure-related hospitalization in the U.S., 1979 to 2004. J Am Coll Cardiol. 2008 Aug 5;52(6):428-34. doi: 10.1016/j.jacc.2008.03.061. PMID 18672162
- [Background] Swank AM, Horton J, Fleg JL, Fonarow GC, Keteyian S, Goldberg L, Wolfel G, Handberg EM, Bensimhon D, Illiou MC, Vest M, Ewald G, Blackburn G, Leifer E, Cooper L, Kraus WE; HF-ACTION Investigators. Modest increase in peak VO2 is related to better clinical outcomes in chronic heart failure patients: results from heart failure and a controlled trial to investigate outcomes of exercise training. Circ Heart Fail. 2012 Sep 1;5(5):579-85. doi: 10.1161/CIRCHEARTFAILURE.111.965186. Epub 2012 Jul 6. PMID 22773109